CLINICAL TRIAL: NCT05027620
Title: Continued Support for Physical Activity in Everyday Life With Parkinson's Disease Using eHealth Technology
Brief Title: Feasibility of Motor-cognitive Home Training for Parkinson's Disease Using eHealth Technology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stiftelsen Stockholms Sjukhem (Other)
Responsible Party: Principal Investigator, Breiffni Leavy, Principal Investigator, Stiftelsen Stockholms Sjukhem
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-03655
Record Dates: First submitted 2021-08-12; First posted 2021-08-30 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-05

CONDITIONS: Idiopathic Parkinson Disease; Telerehabilitation; Physical Therapy
Keywords: Motor-cognitive training; Home training
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Feasibility study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Home training (Experimental): Participants train 3 times weekly in their home environment with help of a digital training app, over a 10-week period.
  Interventions: Other: Motor-cognitive exercise therapy in the home

INTERVENTIONS:
Other: Motor-cognitive exercise therapy in the home — Participants engage in a progressive 10-week exercise program targeted at improving motor and cognitive function. Motor exercises target functional strength, gait and physical activity level. Training sessions occur 3 times weekly and supported by a digital application which has been adapted for people with Parkinson's disease. Weeks 1-2 focus solely on motor exercises. Dual-task (Motor-cognitive) exercises are introduced at week 3 and progressed until week 10. Participants are also encouraged to increase the physical activity levels during the 10 week period.
  Weekly contact is made using the video function/ telephone with clinical specialists/ researchers. Two home visits will occur, the first one week prior to the intervention and at the 5-week period. Participants receive motivational messaging and reminders via the app during the intervention period.

SUMMARY:
The purpose of this study is to test the feasibility of a novel motor-cognitive home training intervention using eHealth technology among people with Parkinson's Disease

ELIGIBILITY:
Inclusion Criteria:

* Neurologist diagnosed Idiopathic PD at least 6 months previous to inclusion.
* Hoehn & Yahr stages I-III
* Stable in anti-Parkinson medications three months prior to inclusion.
* The ability to walk walk independently indoors without a walking aid.
* The ability to walk continually with/without a walking aid for at least 5 minutes.

Exclusion Criteria:

* Cognitive impairment affecting the ability to understand or follow verbal or written instructions (Montreal Cognitive Assessment ≤ 21 points).
* Impaired vision and/or impaired communication which hinders participation.
* Major problems with freezing and/or two or more falls in the month previous to inclusion.
* Other existing neurological/ orthopedic or cardiovascular disease which impedes the performance of unsupervised exercise in the home.
* No internet connection in the home.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-10-05 (Actual); Primary Completion 2022-01-14 (Actual); Study Completion 2022-01-14 (Actual)

PRIMARY OUTCOMES:
Participant satisfaction with the eHealth intervention | 10-week period.
  Participants will rate their satisfaction with using a digital survey following each training session. An average value will be calculated. This will measure the feasibility outcome - Acceptability of the intervention.
Participants perceived intensity of the motor exercises | 10-week period.
  Participants will rate the intensity of the intervention using the Borg Rating of perceived, Exertion Scale (6-20) following each training session. According to this scale, lower numbers signify lower levels of exertion, and higher numbers signify higher levels of exertion. The aim is that participants levels of exertion will lie in the middle range (12-17) This will measure the feasibility outcome - Practicality or Ability to carry out the intervention.
Participants perceived difficulty of the motor-cognitive (dual-task) exercises | 10-week period.
  Participants will rate the difficulty of the dual-task exercises using a 0-10 scale (higher scores = higher degree of difficulty) following each exercise session and scores will be averaged over the study period following. This will measure the feasibility outcome - Suitability of the intervention.
Participants actual use of the eHealth training tool | 10-week period.
  Total time logged in to the digital training app will be derived from system and expressed as a percentage of total recommended intervention time. This will measure the feasibility outcome - Demand of the intervention'.
Total number of adverse events during the training sessions | 10 week period
  Participants will report all adverse events such as falls or other injuries acquired during the training session, during a once weekly telephone interview. This will measure the feasibility outcome Safety.

SECONDARY OUTCOMES:
Habitual physical activity | i) Baseline, pre-intervention. ii) Immediately after the intervention (10-week home training)
  Measured by the ActiGraph accelerometer model GT3X+ (ActiGraph, Pensacola, FL, US) worn on the hip for seven consecutive days
Usual and fast walking speed | i) Baseline, pre-intervention. ii) Immediately after the intervention (10-week home training)
  10 meter walk test at self-selected and fast speeds respectively
Functional capacity as well as dual task gait ability | i) Baseline, pre-intervention. ii) Immediately after the intervention (10-week home training)
  Assessed during the 2 minute walk test (2MWT) in single and dual task conditions
Self-reported walk ability | i) Baseline, pre-intervention. ii) Immediately after the intervention (10-week home training)
  Walk-12 G Questionnaire
Lower extremity function | i) Baseline, pre-intervention. ii) Immediately after the intervention (10-week home training)
  30 second chair stand test
Balance performance | i) Baseline, pre-intervention. ii) Immediately after the intervention (10-week home training)
  Mini Balance Evaluation Systems Test (Mini-BESTest)
Self-reported balance confidence | i) Baseline, pre-intervention. ii) Immediately after the intervention (10-week home training)
  Activity-specific Balance Confidence (ABC) scale
Self-reported difficulties across 8 dimensions of daily living | i) Baseline, pre-intervention. ii) Immediately after the intervention (10-week home training)
  The Parkinson's Disease Questionnaire -39 (PDQ-39)
Exercise self-efficacy | i) Baseline, pre-intervention. ii) Immediately after the intervention (10-week home training)
  Swedish Exercise Self-Efficacy Scale (S-ESES)
Executive Function | i) Baseline, pre-intervention. ii) Immediately after the intervention (10-week home training)
  Attention and psychomotor processing speed will be assessed by the Trail making test (TMT) conditions 2 (letter Sequencing) and 4 (number-Letter Switching (set-shifting)) from Delis-Kaplan Executive Function System (D-KEFS). Results are presented as time in seconds.
Verbal Fluency | i) Baseline, pre-intervention. ii) Immediately after the intervention (10-week home training)
  Verbal function, initiation & task-set switching will be assessed by the Verbal fluency (Letter Fluency, Category Fluency, and Category Switching) from Delis-Kaplan Executive Function System (D-KEFS). Raw scores are converted to scaled scores.

CONTACTS AND LOCATIONS:
Overall Officials: Breiffni Leavy, PhD, Principal Investigator — Stockholms sjukhem and Karolinska Institutet
Locations (1):
- Stockholms Sjukhem, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sedhed J, Johansson H, Andersson N, Akesson E, Kalbe E, Franzen E, Leavy B. Feasibility of a novel eHealth intervention for Parkinson's disease targeting motor-cognitive function in the home. BMC Neurol. 2024 Apr 5;24(1):114. doi: 10.1186/s12883-024-03614-2. PMID 38580913